CLINICAL TRIAL: NCT06501612
Title: Pilot RCT Evaluating Clinical Outcomes of Using Undermyfork Mobile App With Dexcom G7 in a Real-World Community Ambulatory Health Setting
Brief Title: Pilot RCT Evaluating Clinical Outcomes of Using Undermyfork Mobile App With Dexcom G7
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Scripps Whittier Diabetes Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 24-8369
Record Dates: First submitted 2024-07-09; First posted 2024-07-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-01

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes Technology; Diabetes Mobile Application; CGM Monitor
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CGM plus Undermyfork group (Experimental): Participants will be provided continuous glucose monitors (Dexcom G7) to monitor blood glucose for the entire duration of this study (i.e., one new device every 10 days for a total of 2 devices) and will be instructed to use the mobile food diary application. A post-Undermyfork satisfaction qualitative interview will be administered and compensation provided when the CGM is removed and survey completed.
  Interventions: Other: Continuous Glucose Monitor and Undermyfork App
- CGM Only group (Active Comparator): Participants will be provided continuous glucose monitors (Dexcom G7) to monitor blood glucose for the entire duration of this study (i.e., one new device every 10 days for a total of 2 devices).
  Interventions: Other: Continuous Glucose Monitor

INTERVENTIONS:
Other: Continuous Glucose Monitor and Undermyfork App — Participants will be provided two Dexcom G7 sensors to wear during the 20-day intervention period (two 10-day devices). Participants will also be instructed to download and use Undermyfork mobile application where they will have access to their history of their blood glucose responses to their meals in Undermyfork. A randomly selected number of participants in this group will be requested to complete a semi-structured qualitative interview to assess satisfaction with using Undermyfork application immediately following the intervention.
  Arms: CGM plus Undermyfork group
Other: Continuous Glucose Monitor — Participants will be provided two Dexcom G7 sensors to wear during the 20-day intervention period (two 10-day devices).
  Arms: CGM Only group

SUMMARY:
This study aims to determine if adding using a mobile diabetes-related health application with CGM device yields significant benefits, contributing to our understanding of the potential advantages and informing future diabetes care practices. The rationale for testing CGM with Undermyfork in individuals with T2D stems from the potential benefits of real-time glucose monitoring and personalized dietary tracking in improving glycemic control and reducing diabetes-related complications. Unlike standard care, which often involves periodic fingerstick glucose testing and limited dietary guidance, the proposed intervention offers continuous monitoring and tailored dietary insights, thus potentially improving overall diabetes management outcomes. The proposed intervention, therefore, deviates from standard care by integrating mobile health apps into the routine for CGM use, offering a novel avenue for enhanced glycemic monitoring and management.

DETAILED DESCRIPTION:
The current research study seeks to determine the feasibility, acceptability, and effectiveness of using continuous glucose monitors (CGM) with and without a digital food diary (Undermyfork) for CGM naïve individuals with type 2 diabetes (T2D) in a real-world large community health setting. Undermyfork, as a novel digital tool, integrates CGM data with meal tracking, offering users insights into their dietary choices and glucose levels. This innovative approach stems from the rationale that real-time continuous glucose monitoring (CGM) can offer valuable insights into glycemic control, thereby enhancing diabetes self-management. In addition, while the number of free health-related mobile applications continues to increase and underscores the growing interest in leveraging technology to improve health outcomes, there is a limited number of apps that are grounded in evidence. This highlights the importance for clinical testing to evaluate the efficiency and practicality of mobile apps aimed at enhancing health behaviors and outcomes, particularly with diabetes.

This study aims to determine if adding using a mobile diabetes-related health application with CGM device yields significant benefits, contributing to our understanding of the potential advantages and informing future diabetes care practices. The rationale for testing CGM with Undermyfork in individuals with T2D stems from the potential benefits of real-time glucose monitoring and personalized dietary tracking in improving glycemic control and reducing diabetes-related complications. Unlike standard care, which often involves periodic fingerstick glucose testing and limited dietary guidance, the proposed intervention offers continuous monitoring and tailored dietary insights, thus potentially improving overall diabetes management outcomes.

This need for new and effective treatments for T2D motivates the exploration of interventions like the proposed study to integrate easy-to-access mobile technology with CGM. Despite the availability of various diabetes management strategies, optimizing glycemic control remains a challenge. By evaluating the clinical and financial benefits of adding a mobile self-management apps to CGM technology, this study contributes to addressing the unmet needs of individuals who are interested in taking an active role in their health, aiming to advance our understanding of effective and patient-centered diabetes care. The potential outcomes of this research can influence future practices in diabetes management, benefiting individuals with T2D and contributing to the broader landscape of diabetes care.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with type 2 diabetes
* Are on any pills or injectable glucose lowering medication regimen except bolus insulin
* Speak, read, and write in English
* Have A1c between 7.7% and 12.5% in the last 90 days
* Have a cell phone that can download the Dexcom G7 and Undermyfork app

Exclusion Criteria:

* Are on bolus insulin
* Are pregnant
* Are currently participating in another diabetes related study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Average Blood Glucose Level as Measured by HbA1c at Baseline, Day 20, and 4 Months | 4 months
  HbA1c is a person's average blood glucose level over the past three months. This measurement will be collected using lab results provided from healthcare provider. Scores below 7% indicate a healthy HbA1c. Scores above 7% indicate increased risk of diabetes-related complications.

SECONDARY OUTCOMES:
Time in Range (CGM Metric) as Measured by Percentage of Blood Glucose Levels Spent in Target Range at Day 20 | 20 days
  Measures the percentage of time a participant's blood glucose levels stay within the target range using a CGM device throughout the 20-day intervention. Target range is defined as having a blood glucose level between 70 and 180 mg/dL. Thus, percent Time in Range = 100 (Number readings in range (70-180mg/dL)/Total number of readings from CGM). Number of readings will be used in calculation, which scale directly with time.
Time Above Range (CGM Metric) as Measured by Percentage of Blood Glucose Levels Spent Above Target Range at Day 20 | 20 days
  Measures the percentage of time a participant's blood glucose levels exceed the target range using a CGM device throughout the 20-day intervention. Above range is defined as having a blood glucose level above 180 mg/dL. Thus, percent Time Above Range = 100 (Number readings above range (>140mg/dL)/Total number of readings from CGM). Number of readings will be used in calculation, which scale directly with time.
Time Below Range (CGM Metric) as Measured by Percentage of Blood Glucose Levels Spent Below Target Range at Day 20 | 20 days
  Measures the percentage of time a participant's blood glucose levels fall below the target range (usually less than 70 mg/dL) using a CGM device throughout the 20-day intervention. Below range is defined as having a blood glucose level below 70 mg/dL. Thus, percent Time Below Range = 100 (Number readings below range (<70mg/dL)/Total number of readings from CGM). Number of readings will be used in calculation, which scale directly with time.
Frequency of Compliance with Diabetes Self-Care Activities as Measured by the Summary of Diabetes Self Care Activities (SDSCA) Survey at Baseline, Day 20, and 4 Months | 4 months
  The Summary of Diabetes Self Care Activities Survey measures frequency and consistency of diabetes self-care activities during the past 7 days. Possible scores range from 0 (0 Days) to 7 (7 Days). Higher scores indicate better compliance with diabetes self-care.
Severity of Diabetes Distress as Measured by the T2-Diabetes Distress Assessment System, Core Subscale at Baseline, Day 20, and 4 Months | 4 months
  The T2-Diabetes Distress Assessment System, Core Subscale produces a total score to reflect overall emotional distress related to diabetes for individuals with type 2 diabetes. Possible scores range from 1 (Not a Problem) to 5 (A Very Serious Problem) with higher scores indicating higher reported levels of diabetes-related distress.
Severity of Social Determinants of Health as Measured by the Scripps Social Determinants of Health Screening Tool at Baseline, Day 20, and 4 Months | 4 months
  The Social Determinants of Health (SDOH) Screening tool measures the environmental conditions where people are born, live, learn, work, and age that affect a wide range of health and quality-of-life outcomes using 12 items. Possible responses include: Yes, No, Decline to Answer, or Unable to Assess. More "yes" responses indicate more severe environmental conditions affecting health.
Comfortability with Using Mobile Applications as a Health Resource as Measured by Two Likert-type Items at 4 Months | 4 months
  The 2 brief items of this measure examine participants' comfort and perceived skills at using mobile health applications for their health on a scale ranging from (1) not comfortable to (5) very comfortable. Higher scores indicate that participant is more comfortable with using mobile health applications as a health resource. This helps identifying patients with adequate mobile health technology literacy.

OTHER OUTCOMES:
Process Indicators (Adoption): Perceptions of Undermyfork | Immediately following intervention completion
  Results of semi-structured interviews will be qualitatively, descriptively analyzed to reveal perceptions of Undermyfork mobile app, implementation efficacy, challenges, satisfaction, and benefits.
Process Indicators (Adoption): Perceptions and Satisfaction of CGM | Immediately following intervention completion
  Results of brief CGM Satisfaction questionnaire analyzed to reveal perceptions and satisfaction of CGM. Higher scores indicate more satisfaction with CGM use.

CONTACTS AND LOCATIONS:
Overall Officials: Athena Philis-Tsimikas, MD, Principal Investigator — Scripps Health
Locations (1):
- Scripps Whittier Diabetes Institute, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No